CLINICAL TRIAL: NCT03145805
Title: Blood Levels of Bupivacaine in Liver Resection Patients Sited With an Epidural Catheter for Postoperative Pain Control
Brief Title: Bupivacaine Levels in Liver Resection Patients
Status: Completed | Type: Observational
Sponsor: Jessica Burjorjee, MD, FRCPC (Other)
Responsible Party: Sponsor-Investigator, Jessica Burjorjee, MD, FRCPC, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Other Study IDs: ANAE-300-16
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hepatectomy; Analgesia, Epidural
Keywords: blood chemical analysis; bupivacaine; local anesthetic toxicity; Drug-Related Side Effects and Adverse Reactions
MeSH Terms: conditions — Agnosia; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Diagnostic 4 ml blood samples will be drawn from 20 liver resection patients sited with an epidural catheter for 3-5 days of bupivacaine infusion to manage their postoperative pain. Blood will be drawn by phlebotomy with standard of care blood blood-work at 4 time points: preoperatively, upon entry to the post-anesthesia care unit, 2 days postoperatively and then immediately before discontinuation bupivacaine infusion. Blood will be immediately centrifuged by the hospital laboratory and plasma divided into 2 aliquots to be stored at -70 until all samples are collected- at which point they will be shipped to collaborators for analysis of AGP as well as bound and unbound bupivacaine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- liver resection patients: Liver resection patients sited with an epidural catheter for bupivacaine infusion for 3-5 days postoperatively to manage postoperative pain

SUMMARY:
Bupivacaine is a local anesthetic commonly used to manage postoperative pain. Liver resection patients typically have an epidural catheter placed preoperatively through which they receive a continuous infusion of bupivacaine and hydromorphone for up to 5 days postoperatively. The liver metabolizes bupivacaine, and produces proteins that bind with bupivacaine to take it out of circulation and thereby reduce its toxicity. Because a portion of the liver is being removed due to pre-existing liver disease, investigators hypothesize that liver resection patients have an impaired ability to clear bupivacaine from circulation that may increase their susceptibility to bupivacaine toxicity. To assess this, investigators will measure free and bound bupivacaine in liver resection patients postoperatively to determine whether bupivacaine reaches toxic levels. Investigators will also quantify binding protein levels to determine if these levels are reduced after surgery, which could contribute to the elevated bupivacaine levels in these patients. Finally, investigators will monitor patients for signs and symptoms associated with bupivacaine toxicity.

DETAILED DESCRIPTION:
This observational study has been approved for ethical compliance by the Queen's University Health Sciences & Affiliated Teaching Hospitals Research Ethics Board. Following signed informed consent, investigators will collect blood samples from 20 liver resection patients preoperatively and then at 3 different time points after their liver surgery at Kingston General Hospital (upon entry to the post-anesthetic care unit [PACU], on postoperative day 2, and immediately prior to discontinuation of the bupivacaine infusion). These blood draws will occur at the same time as standard of care blood draws. Blood will be centrifuged, and plasma will be stored in duplicate at -70°C until all samples are collected. Samples will be shipped to Centre De Recherche, Centre De Hospitalier, de l'Universitie de Montreal (CHUM) in Montreal, Quebec, Canada, for quantification of free and total bupivacaine as well as AGP. In addition to quantifying circulating bupivacaine and AGP concentrations, investigators will also assess postoperative wound pain on a visual analog scale from 0 to 10, and the presence/absence of local anesthetic toxicity symptoms (tremor, tinnitus, dizziness, blurred vision, hypotension and arrhythmia (including bradycardia).6 These will be assessed as close as possible to the blood collection times (preoperatively, upon arrival to the PACU, on postoperative day 2, and immediately prior to discontinuation of the bupivacaine infusion). Finally, demographic and surgical characteristics will be recorded for all participants.

Inclusion criteria are competent ASA I-IV patients 18 years of age and older scheduled for elective liver resection of at least 3 segments who receive epidural bupivacaine infusion for pain control. Exclusion criteria: pregnancy, renal failure requiring dialysis, sepsis, ejection fraction documented as <15%, taking fluvoxamine or itraconazole, and inability to understand and read English.

Investigators have several outcomes of interest in this study. Of primary interest: plasma concentrations of free and bound bupivacaine and AGP at various time points after surgery. Additional outcomes of interest are pain scores and signs or symptoms of local anesthetic toxicity. Demographic and surgical characteristics will be collected for each patient. Descriptive, univariate and multivariable analyses will be completed with the assistance of a biostatistician.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo elective liver resection surgery
* indicated to be sited with an epidural catheter for bupivacaine infusion for the management of postoperative pain
* competent to provide informed consent
* American anesthesiologists physical classification of I-IV

Exclusion Criteria:

* pregnant
* renal failure requiring dialysis
* sepsis
* ejection fraction documented as <15%
* taking fluvoxamine or itraconazole
* unable to understand or read English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty patients over 18 years of age scheduled to undergo elective liver resection surgery and placement of an epidural catheter for continuous bupivacaine infusion to manage pain for 3-5 days postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
bound bupivacaine levels-1 | 1-2 hours following surgery
  plasma bound bupivacaine levels in liver resection patients upon entry to the post anesthesia care unit
bound bupivacaine levels-2 | 48 hours following surgery
  plasma bound bupivacaine levels on postoperative day 2.
bound bupivacaine levels-3 | 72-120 hours following surgery
  plasma bound bupivacaine levels upon discontinuation of bupivacaine infusion (3-5 days postoperatively)
unbound bupivacaine levels-4 | 1-2 hours following surgery
  plasma unbound bupivacaine levels in liver resection patients upon entry to the post anesthesia care unit
unbound bupivacaine levels-5 | 48 hours following surgery
  plasma unbound bupivacaine levels on postoperative day 2.
unbound bupivacaine levels-6 | 72-120 hours following surgery
  plasma unbound bupivacaine levels upon discontinuation of bupivacaine infusion
alpha-1-acid glycoprotein levels-(AGP)-1 | 1 hour preoperatively
  plasma AGP levels preoperatively
alpha-1-acid glycoprotein levels-(AGP)-2 | 1-2 hours postoperatively
  plasma AGP levels postoperatively upon entry to the post anesthesia care unit
alpha-1-acid glycoprotein levels-(AGP)-3 | 48 hours postoperatively
  plasma AGP levels on postoperative day 2
alpha-1-acid glycoprotein levels-(AGP)-4 | 72-120 hours postoperatively
  plasma AGP levels upon discontinuation of the bupivacaine infusion 3-5 days postoperatively

SECONDARY OUTCOMES:
signs/symptoms of local anesthetic toxicity-1 | 1 hour preoperatively
  tremor, tinnitus, dizziness, blurred vision, hypotension and arrhythmia (including bradycardia)-preoperatively
signs/symptoms of local anesthetic toxicity-2 | 1-2 hours postoperatively
  tremor, tinnitus, dizziness, blurred vision, hypotension and arrhythmia (including bradycardia)-upon entry to the post anesthesia care unit
signs/symptoms of local anesthetic toxicity-3 | 48 hours postoperatively
  tremor, tinnitus, dizziness, blurred vision, hypotension and arrhythmia (including bradycardia)-on postoperative day 2
signs/symptoms of local anesthetic toxicity-4 | 72-120 hours postoperatively
  tremor, tinnitus, dizziness, blurred vision, hypotension and arrhythmia (including bradycardia)-upon discontinuation of bupivacaine infusion-3-5 days postoperatively
surgical site pain-1 | 1 hour preoperatively
  reported pain score of surgical area preoperatively on a scale of 0-10
surgical site pain-2 | 1-2 hours postoperatively
  reported pain score of surgical area preoperatively on a scale of 0-10 upon entry to PACU
surgical site pain-3 | 48 hours postoperatively
  reported pain score of surgical area preoperatively on a scale of 0-10 on postoperative day 2
surgical site pain-4 | 72-120 hours postoperatively
  reported pain score of surgical area preoperatively on a scale of 0-10 upon discontinuation of the bupivacaine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Burjorjee, MD, FRCPC, Principal Investigator — Queen's University/Kingston General Hospital
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burjorjee J, Phelan R, Hopman WM, Ho AM, Nanji S, Jalink D, Mizubuti GB. Plasma bupivacaine levels (total and free/unbound) during epidural infusion in liver resection patients: a prospective, observational study. Reg Anesth Pain Med. 2022 Aug 24:rapm-2022-103683. doi: 10.1136/rapm-2022-103683. Online ahead of print. PMID 36002226